CLINICAL TRIAL: NCT00176540
Title: A Pilot Trial to Evaluate the Effects of Dextromethorphan in Patients Suffering From Cancer-Related Fatigue
Brief Title: Dextromethorphan in Treating Patients With Fatigue Caused by Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Susan Goodin, MD, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000539650; P30CA072720 (NIH); CINJ-5017v2; CINJ-4598; CINJ-NJ11005
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Fatigue; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific; fatigue
MeSH Terms: conditions — Fatigue | interventions — Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dextromethorphan hydrobromide

SUMMARY:
RATIONALE: Dextromethorphan may help relieve fatigue in patients with cancer.

PURPOSE: This clinical trial is studying how well dextromethorphan works in treating patients with fatigue caused by cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the effects of dextromethorphan hydrobromide in patients with cancer-related fatigue.

Secondary

* Correlate the changes in cancer-related fatigue with the levels of plasma homocysteine versus red blood cell folate.

OUTLINE: This is a multicenter, open-label, pilot study.

Patients receive oral dextromethorphan hydrobromide 3 times a day on days 1-7. Treatment repeats weekly for up to 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of malignancy

  * Must be undergoing active treatment for malignancy which may include hormonal therapy (e.g., tamoxifen citrate or leuprolide acetate), but not radiotherapy alone
* Fatigue score ≥ 4 on a verbal analogue scale of 0 to 10
* No untreated cancer-related anemia

PATIENT CHARACTERISTICS:

* Hemoglobin > 10 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow pills
* No known allergy to dextromethorphan hydrobromide
* No patients known to be phenotypically poor metabolizers of CYP2D6
* No untreated hypothyroidism

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior single-dose inhibitors (e.g., ranitidine or cimetidine) for hypersensitivity prophylaxis allowed
* Erythropoietic growth factor therapy of > 8 weeks duration allowed
* No concurrent CYP2D6 inducers or inhibitors
* No concurrent monoamine oxidase inhibitors
* No other concurrent medications containing dextromethorphan hydrobromide
* No concurrent over-the-counter medication, herbal product, vitamin, food supplement, or any other type of special product unless permission to continue use is obtained from the Principal Investigator
* No other concurrent anticancer investigational agents or therapies

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Efficacy

SECONDARY OUTCOMES:
Correlation of the changes in cancer-related fatigue with the levels of plasma homocysteine versus red blood cell folate

CONTACTS AND LOCATIONS:
Overall Officials: Susan Goodin, PharmD, FCCP, BCOP, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/show/NCT00176540